CLINICAL TRIAL: NCT06299995
Title: Cross-sectional, Multicentre and Multidisciplinary Study Describing Phenotype and Burden of a Midfacial Segment Pain
Brief Title: Phenotype and Burden of a Midfacial Segment Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Swiat Zdrowia (Other)
Responsible Party: Principal Investigator, Marcin Straburzynski, Dr, University of Warmia and Mazury in Olsztyn
Other Study IDs: MFSP
Record Dates: First submitted 2024-02-24; First posted 2024-03-08 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Facial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to describe midfacial segment pain phenotype, burden and comorbidities in a multicentre and multidisciplinary setting. The ultimate goal is a comprehensive description of this type of pain allowing for its implementation in future classifications.

This cross-sectional study is designed to describe midfacial segment pain in a clinical setting. Patients from rhinologic, headache and facial pain or oral medicine/dentistry secondary care centres will be recruited during a one year period. Individuals with other facial pain according to current classification such as sinonasal disorders, neoplasms, local infections, history of significant trauma associated with pain onset will be excluded. Data will be collected through a structured questionnaire covering pain characteristics, coexisting diagnoses, pain-related burden and consequences, physical examination and paranasal sinuses imaging.

DETAILED DESCRIPTION:
https://journals.sagepub.com/doi/10.1177/25158163241235642

ELIGIBILITY:
Inclusion criteria

The study will include patients consulting rhinologic, oral medicine/dentistry, headache or pain specialists because of facial pain with the following features:

* located at least partially within an area innervated by the second or third division of the trigeminal nerve (both bilateral and unilateral)
* duration of attacks of > 5 minutes and < 1 month
* attacks recur for > 1 month
* at least one pain-free day per month (this pain-free day must be unrelated to the use of abortive or prophylactic treatment modalities).

Exclusion criteria

1. Facial pain can be attributed to other ICOP-1 diagnosis, apart from tension-type orofacial pain. This means that investigators should exclude especially:

   * facial migraine by ensuring that facial pain is not accompanied by either migraine aura AND/OR nausea/vomiting AND/OR photo- and phonophobia
   * persistent idiopathic facial pain by ensuring that the patient experienced a pain-free day or days in the last month (this day or days must be unrelated to use of abortive or prophylactic treatment modalities).
   * stomatognathic disorders incl. myofascial orofacial pain (chapter 1-3 of ICOP-1) by ensuring that pain is neither unrelated to jaw motion, function or parafunction nor that signs of temporomandibular disorders are present on physical examination.
2. Facial pain with clear rhinogenic cause, such as acute and chronic rhinosinusitis fulfilling both clinical and endoscopic/imaging diagnostic criteria according to the European Position Paper on Rhinosinusitis and Nasal Polyps (EPOS 2020).
3. Facial pain that can be attributed to neoplasms.
4. Facial pain that can be attributed to local infection including post-herpetic neuralgia.
5. History of significant trauma associated with pain onset (pain developed within 7 days from trauma).

Patients who additionally and independently suffer from primary headaches whose mid-facial pain cannot be explained as orofacial headaches are explicitly not excluded. In other words, patients with migraine are not excluded, as long as their facial pain has no typical migraine features (i.e. nausea/vomiting, photo- AND phonophobia or aura) and facial pain attacks occur independently of headache episodes.

Also, patients showing signs of mucosal contact points or deviated nasal septum will be included, but the presence of these conditions should be noted in the patients' history. Moreover, patients with Lund-Mackay score of 4 or less can be included in the study, unless any singular sinus can be scored with 2 points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting rhinologic, dentistry, headache or pain specialists because of facial pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain characteristics | 1 month prior to study visit.
  Following pain features will be assessed with structured questionnaire: location, frequency, duration, quality, intensity, accompanying symptoms, provoking/relieving factors.

SECONDARY OUTCOMES:
Coexisting diagnoses | 1 month prior to study visit.
  Other headache/pain-related disorders (assessed with structured questionnaire).
Pain-related burden and consequences | 1 month prior to study visit.
  Medications used and their efficacy, consultations in the past, surgical procedures in the past, cost of treatment (assessed with structured questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Straburzyński, PhD, Principal Investigator — University of Warmia and Mazury in Olsztyn
Locations (13):
- Department of Otolaryngology, University of Malta, Msida, Malta
- Poland (10):
  - Athleticomed - Pain&Headache Treatment Centre, Bydgoszcz
  - Department of Otolaryngology, Head and Neck Surgery and Laryngological Oncology, Bydgoszcz
  - Department of Neurology, Jagiellonian University Medical College, Krakow
  - Świat Zdrowia, Orzyny
  - Department of Neurology and Restorative Medicine, Health Institute dr Boczarska-Jedynak, Oświęcim
  - 4. Department of Otorhinolaryngology, National Institute of Medicine of the Ministry of the Interior and Administration, Warsaw
  - 5. Department of Otolaryngology, Centre of Postgraduate Medical Education, Warsaw
  - Department of Experimental Dentistry, Wroclaw Medical University, Wroclaw
  - Department of Neurology, Wroclaw Medical University, Wroclaw
  - MIGRE Polish Migraine Center, Wroclaw
- United Kingdom (2):
  - Pain Medicine, Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Department of Otorhinolaryngology, Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No